CLINICAL TRIAL: NCT04326114
Title: Effectiveness and Safety of Respiratory Training Devices in the Prevention and Severity of COVID-19: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness and Safety of Respiratory Training in the Prevention and Severity of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Covid_ISCIII 20/265-E_BS
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Disease, Infectious; Respiratory Disease; Safety Issues; Effectiveness
MeSH Terms: conditions — Communicable Diseases; Respiration Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory training (Experimental)
  Interventions: Device: Inspiratory training device
- Expiratory training (Experimental)
  Interventions: Device: Expiratory training device
- Control (No Intervention)

INTERVENTIONS:
Device: Inspiratory training device — Inspiratory training by a Power-breath device
  Arms: Inspiratory training
Device: Expiratory training device — Expiratory training a Winner-flow device
  Arms: Expiratory training

SUMMARY:
A randomized controlled clinical trial will be carried out using inspiratory and expiratory training devices on healthy subjects recruited in social networks and university environments. The aim will be to determine the effectiveness and safety in the prevention and severity of COVID-19 disease by a respiratory training with inspiratory and expiratory devices.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Drugs
* Surgery
* Neurology diseases
* Rheumatic diseases
* Systemic diseases
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-07-26 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
COVID-19 disease diagnosis | Change from Baseline COVID-19 disease diagnosis at 8 weeks
  Dichotomous categorical variable measured by "yes" or "no" responses

SECONDARY OUTCOMES:
COVID-19 disease symptoms severity | Change from Baseline COVID-19 disease symptoms severity at 8 weeks
  Dichotomous categorical variable measured by "slight" or "severe" responses
Adverse effects | Change from Baseline adverse effects at 8 weeks
  Polytomous categorical variable measured by adverse effects responses

IPD SHARING:
Plan to Share IPD: No